CLINICAL TRIAL: NCT05654129
Title: Non-interventional Study Exploring the Relationship Between Porphyromonas Gingivalis and the Severity of Fibrosis in Patients With Non-alcoholic Fatty Liver Disease (NAFLD)
Brief Title: Porphyromonas Gingivalis and Severity of Fibrosis in Patients With Non-alcoholic Fatty Liver Disease
Acronym: BUCCONAFLD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RC31/19/0043
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: people with stage F1-F2 NAFLD versus people with stage F3-F4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F1-F2 NAFLD (Other): Patients with NAFLD stage 1 or 2 confirmed by a biopsy less than 1 year old
  Interventions: Other: saliva samples; Other: medical questionnaire
- F3-F4 NAFLD (Other): Patients with NAFLD stage 3 or 4 confirmed by a biopsy less than 1 year old
  Interventions: Other: saliva samples; Other: medical questionnaire

INTERVENTIONS:
Other: saliva samples — saliva samples (non-invasive, in the sites evaluated during the partial survey) will be perform by one of the investigators .
Other: medical questionnaire — a complete medical questionnaire will be carried out (general, lifestyle and quality of life) will be perform by one of the investigators .

SUMMARY:
Many studies suggest that Porphyromonas gingivalis, a virulent periodontopathogenic bacterium, is associated with many systemic diseases such as cardiovascular diseases. In addition, a recent study showed the impact of Porphyromonas gingivalis on Non-Alcoholic Steatosis Liver Disease (NASH). It would be responsible for aggravation of non-alcoholic fatty liver disease (NAFLD) by stimulating inflammation in the damaged liver tissue.

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease is becoming the leading cause of chronic liver disease with a prevalence of 20% worldwide. The prognosis depends on the degree of fibrosis: patients with a low degree of fibrosis (F0-F2) have a good prognosis unlike those with severe fibrosis or cirrhosis (F3-F4), exposed to excess mortality from cardiovascular diseases , cancers, and complications of cirrhosis. The diagnosis of the fibrosis stage is histological but the worsening of the fibrosis remains unknown.

The intestinal microbiota is an etiological factor in NAFLD and dysbiosis is associated with the severity of fibrosis. There is also a physiopathological rationale between oral bacterial microbiota and NAFLD. The oral microbiota is very rich, it corresponds to a reservoir of 1010 bacteria of Gram-negative bacteria (BGN). Its dysbiosis causes oral infections like periodontal diseases, immuno-infectious pathologies linked to an imbalance between the bacterial etiological factor and the host's immune defenses.

Many studies suggest that Porphyromonas gingivalis, a virulent periodontopathogenic bacterium, is associated with many systemic diseases such as cardiovascular diseases. In addition, a recent study showed the impact of Porphyromonas gingivalis on Non-Alcoholic Steatosis Liver Disease (NASH). It would be responsible for aggravation of non-alcoholic fatty liver disease (NAFLD) by stimulating inflammation in the damaged liver tissue.

the hypothesis that the salivary levels of Porphyromonas Gingivalis could be associated with the degree of severity of fibrosis in NAFLD patients, and would constitute a new therapeutic target for the evaluation of fibrosis. This work would open new perspectives in treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* subjects with NAFLD confirmed by a biopsy less than 1 year old
* subjects over the age of 18
* subjects able to receive information on the course of the study and to understand the information form to participate in the study
* the subjects who gave their non-objection to participate in the study

Exclusion Criteria:

* Having another associated cause of liver disease or steatosis such as viral infections and autoimmune disease
* With alcohol consumption >30g/d (men) or 20g/d (women)
* With a history of cirrhosis decompensation
* Having taken antibiotics, prebiotics or probiotics in the month prior to inclusion
* With chronic or acute gastrointestinal disease
* With a history of gastrointestinal surgery modifying the anatomy
* During pregnancy or breastfeeding
* With a history of oral surgery in the month prior to inclusion
* For whom oral surgery is planned between the collection of the non-objection and the inclusion in the odontology service
* At risk of infection (existence of one or more known chronic infectious pathologies) and/or chronic renal failure (creatinine clearance < 60ml/min).
* Suffering from a general pathology contraindicating the performance of diagnostic procedures such as periodontal probing (patients at high risk of infective endocarditis according to the French National Agency for the Safety of Medicines and Health Products ANSM)
* Under legal protection, dependent, under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2023-12-05 (Estimated)

PRIMARY OUTCOMES:
frequency of Porphyromonas gingivalis in the saliva | 1 day
  compare the mean frequency of Porphyromonas gingivalis in the saliva of people with stage F1-F2 NAFLD versus people with stage F3-F4.

CONTACTS AND LOCATIONS:
Overall Officials: Vincent BLASCO-BAQUE, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU Toulouse, Toulouse, France

IPD SHARING:
Plan to Share IPD: No